CLINICAL TRIAL: NCT05982756
Title: A Prospective Randomized Controlled Clinical Study of Bortezomib Combined With DAG Regimen in the Treatment of Refractory/Relapsed AML
Brief Title: Bortezomib Combined With DAG Regimen in the Treatment of Refractory/Relapsed AML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04
Record Dates: First submitted 2023-07-13; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-03

CONDITIONS: Bortezomib; Acute Myeloid Leukemia
Keywords: pre-excitation regimen; acute myeloid leukemi; Bortezomib
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Bortezomib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Remove masking if necessary
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group: Induction treatment plan A (Experimental): Bortezomib+DAG pre-excitation regimen
  Interventions: Drug: DAG pre-excitation regimen with Bortezomib
- Control group: induction regimen B (Active Comparator): DAG pre-excitation plan alone
  Interventions: Drug: DAG pre-excitation regimen with Bortezomib

INTERVENTIONS:
Drug: DAG pre-excitation regimen with Bortezomib — Bortezomib+DAG pre-excitation regimen: Bortezomib (specification 3.5mg, intravenous injection, 4 times a course of treatment, 1.3mg/m2, d1, 4, 8, 11; doxorubicin liposome injection 5 mg/ m2, intravenous infusion, once every other day, 5 times in total; cytarabine 10 mg/m2 every 12 hours, subcutaneous injection, d1-14; G-CSF 200 μg/m2 daily, subcutaneous injection, d1-14 Days, WBC >10×109/L during chemotherapy, postpone the use until it falls below this value;
  Other Names: Bortezomib group

SUMMARY:
In recent years, the efficacy of AML has been greatly improved, which is mainly due to the following aspects: the development of individualized treatment strategies based on genetic prognosis stratification, the application of high-dose cytarabine-containing induction and consolidation regimens , the choice of allogeneic or autologous hematopoietic stem cell transplantation, etc. However, 20%-30% of young patients and 40%-50% of elderly patients will relapse again, and 20%-40% of patients cannot be relieved after standard induction regimens, that is, relapsed and refractory AML. The re-induction remission rate is low, the survival period is short, and the prognosis is extremely poor. There is still a lack of standard treatment options. Although a small number of patients can benefit from allogeneic hematopoietic stem cell transplantation (allo-HSCT), most patients lack suitable donors. The choice of high-dose chemotherapy is a salvage treatment option, but treatment-related hematological or non-hematological toxicities and high lethality make the option controversial, especially for the elderly. The development of new low-toxic targeted drugs is a future trend, and the design of new efficient and safe chemotherapy regimens is also a way of thinking. This study designed a prospective single-center clinical randomized controlled study plan, that is, the use of bortezomib (1.3mg/m2, d1, 4, 8, 11) combined with DAG regimen in the treatment of refractory/relapsed AML, to evaluate the clinical efficacy (complete remission rate , total effective rate, 2-year progression-free survival rate and 2-year overall survival rate), and observe how safe the new program is. The results of the research will make it possible to design a high-efficiency, low-toxicity and high-feasibility chemotherapy regimen for refractory/relapsed patients, and guide the clinical treatment of relapsed/refractory acute leukemia.

DETAILED DESCRIPTION:
This study aimed to evaluate the clinical efficacy of bortezomib combined with DAG regimen in the treatment of refractory and relapsed AML (complete remission rate, overall effective rate, 2-year progression-free survival rate and 2-year overall survival rate), and to compare the effects of the two regimens. Safety, guiding the clinical treatment of relapsed/refractory acute leukemia. For the smooth development of this study, the relevant monitoring indicators of the study are as follows:

1. Select suitable subjects with relapsed/refractory acute myeloid leukemia according to the inclusion criteria, and explain the treatment indications of bortezomib and the purpose of this clinical study to the subjects and their families.
2. The attending doctor communicates with the subject and his family members according to the condition of the subject and signs the informed consent. The subject needs to perform the following tests: three routine tests, cerebrospinal fluid routine and biochemistry, liver function, kidney function, PNH test, anemia four Items (ferritin, folic acid, vitamin B12, erythropoietin), blood sugar, blood lipids, electrolytes, myocardial enzymes, coagulation function, HIV antibody, syphilis, screening of related hepatitis virus markers, tumor markers, chest X-ray, Electrocardiogram, CT or MRI examination, etc.; if conditions permit, immune function and T cell subsets can be monitored.
3. Clinical research: According to the research design, this clinical research was carried out, and relevant indicators such as the incidence of third-degree and fourth-degree myelosuppression and infection after chemotherapy, the rate of antibiotic use, the delay rate of chemotherapy, and the extension time of chemotherapy were recorded. The incidence and severity of adverse drug reactions were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with AML confirmed by bone marrow morphology and immunology
2. Patients who do not respond or relapse after conventional treatment
3. Age 18-75
4. Liver and kidney function: blood bilirubin ≤ 35 μmol/L, AST/ALT below 2 times the upper limit of normal value, 451 μmol/L ≥ serum creatinine ≥ 133 μmol/L, 80 ml/min ≥ creatinine clearance ≥ 20ml/min
5. Cardiac function index EF value ≥ 50%
6. Physical condition score 0-2 (ECOG score)
7. Obtain signed informed consent from patients or family members

Exclusion Criteria:

1. Allergies or obvious contraindications to any of the drugs involved in the program
2. Severe heart disease, including myocardial infarction and cardiac insufficiency.
3. Suffering from other organ malignancies at the same time
4. Active tuberculosis patients and HIV positive patients
5. Suffering from other blood system diseases at the same time
6. Pregnant or lactating women
7. Inability to understand or follow the research protocol

1. Past history of intolerance or allergy to similar drugs 2. Patients under 18 years old or over 75 years old 3. Simultaneously participate in other clinical investigators 4. Any other circumstances that prevent the conduct of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate Rate of bone marrow blasts | Evaluation at the 4th weekend after the end of all chemotherapy cycles
  Bone marrow blasts <20%

SECONDARY OUTCOMES:
blood routine | Evaluation at the 4th weekend after the end of all chemotherapy cycles
  differential blood count
liver function | Evaluation at the 4th weekend after the end of all chemotherapy cycles
  Detection of hepatic metabolite concentration in blood
Recovery time | Evaluation at the 4th weekend after the end of all chemotherapy cycles
  Recovery time of patients' neutrophils, hemoglobin and platelets
The incidence of complications in patients | Evaluation at the 4th weekend after the end of all chemotherapy cycles
  The incidence of complications in patients
kidney function | Evaluation at the 4th weekend after the end of all chemotherapy cycles
  Urine composition analysis

CONTACTS AND LOCATIONS:
Overall Officials: Fuling Zhou, phD, Study Director — Wuhan University; TIANZHI WU, phD, Principal Investigator — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China